CLINICAL TRIAL: NCT06909734
Title: Trauma-Informed Motivational Interviewing as a Frontrunner Paradigm for Addressing Leprosy-Related Discrimination, Body Image Dissatisfaction, Resilience, and Social Engagement in Rural Dwelling Samples
Brief Title: Trauma-Informed Motivational Interviewing in Rural Dwelling Samples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, Rasha Eweida, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2232025
Record Dates: First submitted 2025-03-22; First posted 2025-04-03 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Discrimination, Perceived
Keywords: Leprosy; Discrimination; Body Image; Resilience; Social
MeSH Terms: conditions — Perceived Discrimination; Leprosy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- interventional group (Experimental): This investigation will draw upon existing literature exploring the intersection of TIMI in Leprosy-Related Discrimination, Body Image Dissatisfaction, Resilience, and Social Engagement in Rural Dwelling Samples. By understanding how Threat to Identity and Meaning in Illness (TIMI) influences the psychological and social impact of leprosy-related discrimination. It explores how body image dissatisfaction affects self-perception and mental health while assessing resilience as a coping mechanism. Additionally, it examines social engagement in rural settings, where stigma may lead to isolation. The findings can inform targeted mental health interventions and stigma-reduction strategies to support affected individuals.
  Interventions: Behavioral: Trauma-Informed Motivational Interviewing
- control group (Placebo Comparator): traditional standardized care such as Group Therapy/ peer support.
  Interventions: Behavioral: Trauma-Informed Motivational Interviewing

INTERVENTIONS:
Behavioral: Trauma-Informed Motivational Interviewing — Trauma-Informed Motivational Interviewing: Core Principles
  TIMI integrates two evidence-based approaches: Trauma-Informed Care (TIC) and Motivational Interviewing (MI). TIC emphasises understanding and acknowledging the impact of trauma on individuals' behaviours and emotional well-being. MI, a client-centred approach, fosters intrinsic motivation for change by exploring ambivalence and strengthening personal autonomy.

SUMMARY:
Leprosy remains a profoundly stigmatized condition in many rural communities worldwide, fostering social exclusion, body image dissatisfaction, and diminished mental health outcomes. TTrauma-Informed Motivational Interviewing (TIMI) emerges as a promising paradigm to address these psychosocial challenges, enhancing resilience, improving self-perception, and fostering social re-engagement.

DETAILED DESCRIPTION:
Introduction

Leprosy remains a profoundly stigmatised condition in many rural communities worldwide, fostering social exclusion, body image dissatisfaction, and diminished mental health outcomes. Traditional biomedical approaches, while essential for physical recovery, often neglect the psychological and social ramifications of the disease. Trauma-Informed Motivational Interviewing (TIMI) emerges as a promising paradigm to address these psychosocial challenges, enhancing resilience, improving self-perception, and fostering social re-engagement.

Understanding the Psychological Impact of Leprosy

Leprosy-related stigma is multifaceted, rooted in cultural beliefs, misinformation, and visible physical impairments. Affected individuals frequently endure social rejection, which fosters feelings of shame, body image dissatisfaction, and emotional distress. These experiences, akin to trauma, may disrupt self-efficacy and hinder engagement with both healthcare systems and social networks.

Trauma-Informed Motivational Interviewing: Core Principles

TIMI integrates two evidence-based approaches: Trauma-Informed Care (TIC) and Motivational Interviewing (MI). TIC emphasises understanding and acknowledging the impact of trauma on individuals' behaviours and emotional well-being. MI, a client-centred approach, fosters intrinsic motivation for change by exploring ambivalence and strengthening personal autonomy.

The synergy of TIMI rests on five core principles:

Safety: Ensuring physical and emotional safety in all interactions.

Trustworthiness and Transparency: Building a collaborative, open relationship.

Peer Support and Empowerment: Encouraging individuals to harness personal and community strengths.

Collaboration and Mutuality: Shifting the power dynamic to promote shared decision-making.

Cultural, Historical, and Gender Awareness: Respecting cultural narratives and addressing systemic inequalities.

Addressing Key Psychosocial Challenges

Combatting Discrimination and Stigma: TIMI helps reframe self-perceptions, encouraging individuals to challenge internalised stigma and societal bias. By fostering empathy and understanding, community members may also engage in reducing discriminatory attitudes.

Improving Body Image and Self-Esteem: Acknowledging the emotional weight of physical changes, TIMI supports individuals in developing healthier self-concepts. Through guided dialogue, participants explore their strengths and redefine their value beyond appearance.

Building Resilience: TIMI fosters a growth mindset, promoting coping strategies that empower individuals to navigate adversity. This is crucial in rural settings where access to mental health services may be limited.

Enhancing Social Engagement: By empowering participants to explore their personal goals and values, TIMI helps identify pathways to meaningful social connections, promoting reintegration into community life.

Implementation in Rural Contexts

Adapting TIMI to rural environments necessitates a culturally sensitive approach. Training local healthcare providers, community leaders, and peer mentors in TIMI principles ensures sustainability. Additionally, integrating TIMI within existing community health frameworks, such as primary healthcare clinics or local support groups, facilitates accessibility.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a confirmed medical diagnosis of leprosy (current or past) experiencing physical, emotional, or social consequences.

Exclusion Criteria:

* Severe Cognitive or Psychiatric Impairments:

Individuals with severe mental health conditions (e.g., untreated psychosis, severe intellectual disabilities) that impede the reflective, goal-setting nature of Motivational Interviewing.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Leprosy-Related Discrimination | 1 month and half
  To assess the stigma surrounding leprosy, this scale comprises four domains: Experienced stigma, Disclosure concerns, Internalized stigma, and Anticipated stigma. Each domain aims to capture different facets of the stigma experienced by individuals affected by leprosy. With a total of 21 questions, the SARI Stigma Scale explores how patients encounter stigma in their daily lives. The scoring method used is that if the patient answers no, do not know, or it is not relevant, they will be given a score of zero, whereas if they answer yes, the patient will receive a score ranging from one to three depending on the frequency the patient experiences.

SECONDARY OUTCOMES:
Body Image Psychological Inflexibility Scale (BIPIS). | 1 month and half
  Body Image Psychological Inflexibility Scale (BIPIS). The BIPIS was developed by the Callaghan et al., (2015) and is the scale under investigation. The tool resulted in 16-item scale had high internal consistency (%0.93). Scores on the BIPIS are calculated by summing the total (item 9 is reverse scored); higher scores indicate greater psychological inflexibility. Each item is rated on a Likert-type scale ranging from 1 (never true) to 7 (always true). All BIPIS items are summed for a total, and higher scores are indicative of higher levels of psychological inflexibility in body image.

CONTACTS AND LOCATIONS:
Overall Officials: rasha eweida, Principal Investigator — Alexandria University
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No